CLINICAL TRIAL: NCT04411771
Title: Evaluation of PCBH in Primary Care With or Without Additions of Guided Self-help CBT - a Single-blind Randomised Clinical Trial and Preparation for a Multi-center Study
Brief Title: PCBH With the Addition of Self-help CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Kronoberg County Council (Other Government); Capio Group (Other)
Responsible Party: Principal Investigator, Viktor Kaldo, Professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00699
Record Dates: First submitted 2020-05-06; First posted 2020-06-02 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Depression, Anxiety; Quality of Life; Psychological Distress; Activities, Daily Living; Insomnia; Stress
Keywords: PCBH; Primary Care Behavioral Health; Integrated Behavioural Health; Primary Care Mental Health Services; Primary Care; Brief Interventions; Focused Acceptance and Commitment Therapy; Brief CBT; IBH; CBT; Self-help; Guided Self-help
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Crisis Intervention; Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Patients are randomised between an extended assessment and a screening assessment. Patients in the screening assessment arm can only be treated with brief interventions whereas patients in the extended assessment arm are offered guided self-help if deemed appropriate and otherwise gets brief interventions.
  Patients are thus randomized to two arms, however we have included four arms in order to be able to describe the primary and secondary analysis. The primary is performed on all patients treated with shCBT in the arm where an extended assessment is made, compared to patients in the screening assessment arm that is found suitable for shCBT (base on screening data), but treated with brief interventions.
Who Masked: Participant
Masking Description: Patients will be informed only that they will be randomised between two different types of extended assessments, both of which are more extensive than regular healthcare. They will receive no information about the nature of the extended assessments or about different treatments following the assessments to avoid nocebo effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Extended Assessment - Given shCBT (Experimental): The extended assessment includes screening instruments, a structured interpretation of the screening instruments, a structured interview and a medical anamnesis. If deemed appropriate, the patient can be offered treatment with guided self help. If the patient's problem is not deemed appropriate for this type of care or if the patient is not interested in guided self-help, they are offered brief interventions (BI).
  In the primary analysis, only patients given shCBT are included
  Interventions: Behavioral: Guided self-help CBT
- Screening Assessment - Suitable for shCBT but given BI (Active Comparator): The screening assessment includes screening instruments and a contextual interview. Patients in this arm will always be treated with brief interventions.
  In the primary anaysis, only patients suited for shCBT are included, as decided from an algorithm based on data from their screening.
  Interventions: Behavioral: Brief interventions
- Extended Assessment - All patients (Experimental): Same as the other arm marked as "Experimental", but for the purpose of a secondary analysis all patients randomized to Extended Assessment are included, regardless of if they start shCBT or BI
  Interventions: Behavioral: Brief interventions; Behavioral: Guided self-help CBT
- Screening Assessment - All patients (Active Comparator): Same as the other arm marked as "Active comparator", but for the purpose of a secondary analysis all patients randomized to Screening Assessment are included, regardless of if they are suiteble for shCBT or not.
  Interventions: Behavioral: Brief interventions

INTERVENTIONS:
Behavioral: Brief interventions — 'Brief Interventions' (BI) is a generic term for a multitude of tools and interventions used in patient visits within PCBH. BI start immediately at the initial consultation, which ends with a personally tailored and evidence-informed plan adjusted to the patient's context. As such, there is no separation between assessment and intervention. The interventions within BI often have their foundation in CBT, ACT or MI. The common theme is that they are principle-based rather than manual-based and focus on behavioral change in relation to a problem that is perceived both possible to affect and relevant to the patient, rather than focusing on a specific diagnosis or condition. Follow-up appointments are scheduled flexibly depending on the patient's perceived need. Usually a BI treatment consists of 1-4 appointments with several weeks apart and ends when the patient feels that they are moving in the right direction.
  Other Names: Focused interventions, brief CBT, focused Acceptance and Commitment Therapy, FACT, focused ACT
  Arms: Extended Assessment - All patients; Screening Assessment - All patients; Screening Assessment - Suitable for shCBT but given BI
Behavioral: Guided self-help CBT — The patient receives a previously scientifically evaluated CBT-based self-help book for one of the following conditions: depression, generalized anxiety disorder, panic disorder, social anxiety, health anxiety, insomnia, or stress/burnout. The therapist support consists of 3-6 contacts throughout the 6-12 weeks long intervention period as decided by the clinician and patient together, as long as at least one and not more than three are physical visits at the center and the rest via phone, video conferencing, or secure internet messages. Clinicians delivering shCBT will need four days of reading and two days of training to be able to make initial assessments and problem profiling and use the self-help books.
  Other Names: Self-help books, bibliotherapy, self-help CBT
  Arms: Extended Assessment - All patients; Extended Assessment - Given shCBT

SUMMARY:
The overarching goal of primary care is to offer all patients individualized and context-sensitive healthcare with high access and continuity. One of the reasons primary care struggles with this goal is that many patients suffer from mental health problems, while there is a lack of psychosocial resources as well as clear pathways for these patients.

Primary care behavioural health (PCBH, in Swedish IBH) is an innovative way of organizing primary care, where psychosocial resources have more and shorter visits, strive for same-day access, and have an active consulting role in the primary care team. To help patients with achieving relevant behavior changes, so called Brief Interventions are used. However, these interventions have not been systematically evaluated in the same way that CBT has, and there is a risk that patients that would have benefitted from structured CBT are undertreated.

This study is a pilot study preparing for a large multicenter study that will be conducted starting in late 2020. The investigators want to find out if an addition of an extended evaluation and possibility of treatment with guided CBT self-help can increase the treatment effects of PCBH on patient functioning and symptoms, compared to standard PCBH with a contextual assessment and brief interventions. In the process, the investigators are also conducting one of the first RCT on brief interventions. As this is a pilot study, the feasibility of implementing the study protocol in regular healthcare is also tested in order to collect high-quality data while creating minimal disturbance in the centers' ordinary routines.

PCBH has the potential to increase the quality of care for patients with mental health problems. This study is the first to step towards answering the question if the effects of brief intervention are large enough to merit large-scale implementation, and if an add-on of other brief and easily implemented treatments can increase them.

DETAILED DESCRIPTION:
The overarching goal of primary care is to offer all patients individualized and context-sensitive healthcare with high access and continuity. One of the reasons primary care struggles with this goal is that many patients suffer from mental health problems, while there is a lack of psychosocial resources as well as clear pathways for these patients.

Primary care behavioural health (PCBH, in Swedish IBH) is an innovative way of organizing primary care, where psychosocial resources have more and shorter visits, strive for same-day access, and have an active consulting role in the primary care team. To help patients with achieving relevant behavior changes, so called Brief Interventions are used. However, these interventions have not been systematically evaluated in the same way that CBT has, and there is a risk that patients that would have benefitted from structured CBT are undertreated.

This study is a pilot study preparing for a large multicenter study that will be conducted starting in late 2020. The investigators want to find out if an addition of an extended evaluation and possibility of treatment with guided CBT self-help can increase the treatment effects of PCBH on patient functioning and symptoms, compared to standard PCBH with a contextual assessment and brief interventions. In the process, the investigators are also conducting one of the first RCT on brief interventions. As this is a pilot study, the feasibility of implementing the study protocol in regular healthcare is also tested in order to collect high-quality data while creating minimal disturbance in the centers' ordinary routines.

Our main research questions are:

1. Does an extended version of PCBH, including an additional assessment and the option of guided self-help CBT when indicated by a patient's problem profile, lead to superior patient outcomes compared to standard PCBH where a brief, contextual assessment followed by Brief Interventions is the only option? If not, can standard PCBH be shown to be non-inferior?
2. Does the addition of guided self-help CBT have a negative effect on availability, reach, and cost-effectiveness compared to standard PCBH? If not, can guided self-help CBT be shown to be non-inferior to standard PCBH concerning these outcomes?

The project is a joint effort by Karolinska Institutet, Linnaeus University, and Capio Närsjukvård and will be conducted as a single-blind (patients) randomized trial within regular healthcare at two primary care centres with a total of approximately 75 patients. Time-points for measures are screening at the initial visit and follow-ups 4, 8 and 52 weeks later. Primary outcome will be the 12-item version of the WHO Disability Assessment Schedule 2.0 (WHODAS-12). This is a condition-independent measure of everyday functioning that has been found to be relevant to mental health.

PCBH has the potential to increase the quality of care for patients with mental health problems. This study is the first to step towards answering the question if the effects of brief intervention are large enough to merit large-scale implementation, and if an add-on of other brief and easily implemented treatments can increase them. Our study will also answer whether the effects can be increased by adding previously empirically supported self-help, while still being cost-effective and maintain high availability of services. The goal is to create a more solid empirical base that can guide decision makers when they balance treatment effects, availability, and costs in determining which organizational models and interventions that are best used in primary care.

If the results are positive, this project functions as a concrete start to a large-scale implementation of this new method, since it is firmly placed within regular primary care and uses highly implementable interventions.

ELIGIBILITY:
Inclusion Criteria:

* All patients from age 18 deemed to be suitable for Behavioral Health interventions, according to screening methods and/or clinical assessments made by health care personnel at the PCC, will be included. This broad criteria reflects the naturalistic setting where decisions of clinicians, rather than highly standardized criteria, are the basis for inclusion.

Exclusion Criteria:

* Does not speak Swedish well enough to fill out questionnaires.
* Is in need of emergency type care, like with suicidal ideation or behaviours, ongoing psychosis or mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
WHO Disability Assessment Schedule 2.0 12-item (WHODAS-12) (4 domains) | Change during the period Pre-Week4-Week8
  The four domains of Life activities, Cognition, Getting along, and Participation. In the 12-item version of the WHO Disability Assessment Schedule 2.0 (WHODAS-12) will be used as primary outcome, since these are condition-independent measures of Behavioral Health relevant everyday functioning. The scale ranges from 0 to 32 points. A lower score means better functioning. As such, a lower score is a better outcome.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule 2.0 12-item (WHODAS-12) (whole instrument) | Change during the period Pre-Week4-Week8-Week 52
  The two domains of Mobility and Self-care will be measured and the whole WHODAS will be used in some secondary analyses, but not for the primary outcome since these domains tend to form two independent factors, many patients will have initial adequate function in these domains and they are not expected to change much. The scale ranges from 0 to 48 points. A lower score means better functioning. As such, a lower score is a better outcome.
Patient Health Questionnaire 2-Item (PHQ-2) | Change during the period Pre-Week4-Week8-Week 52
  Depressive symptoms are measured with a very short version of a well established patient-rated scale for depression. The scale ranges from 0 to 6 points. A lower score means less depressive symptoms. As such, a lower score is a better outcome.
Generalized Anxiety Disorder 2-Item (GAD-2) | Change during the period Pre-Week4-Week8-Week 52
  Anxiety and worry symptoms are measured with a very short version of a well established patient-rated scale for generalized anxiety disorder. The scale ranges from 0 to 6 points. A lower score means less anxiety and worry symptoms. As such, a lower score is a better outcome.
Social Phobia Inventory - Abbreviated version (Mini-SPIN) | Change during the period Pre-Week4-Week8-Week 52
  Social anxiety symptoms are measured with a very short version of a well established patient-rated scale for social phobia. The scale ranges from 0 to 12 points. A lower score means less symptoms of social anxiety. As such, a lower score is a better outcome.
The Alcohol Use Disorders Identification Test-Concise (AUDIT-C) | Change during the period Pre-Week4-Week8-Week 52
  Symptoms of alcohol misuse are measured with a very short version of a well established patient-rated scale for alcohol misuse. The scale ranges from 0 to 12 points. A lower score means less symptoms of alcohol misuse. As such, a lower score is a better outcome.
Panic Disorder Severity Scale - Self rated 2-item (PDSS-SR-MINI-2) | Change during the period Pre-Week4-Week8-Week 52
  Symptoms of panic attacks are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 8 points. A lower score means less symptoms of panic disorder. As such, a lower score is a better outcome.
Shirom-Melamed Burnout Questionnaire 2-item (SMBQ-MINI-2) | Change during the period Pre-Week4-Week8-Week 52
  Burnout symptoms are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 2 to 14 points. A lower score means less symptoms of burnout. As such, a lower score is a better outcome.
Perceived Stress Scale (PSS-MINI-2) | Change during the period Pre-Week4-Week8-Week 52
  Stress symptoms are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 8 points. A lower score means less stress symptoms. As such, a lower score is a better outcome.
Insomnia Severity Index 2-item (ISI-MINI-2) | Change during the period Pre-Week4-Week8-Week 52
  Symptoms of sleep disorders are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 8 points. A lower score means less sleep problems. As such, a lower score is a better outcome.
Short Health Anxiety Inventory 3-item (SHAI-MINI-3) | Change during the period Pre-Week4-Week8-Week 52
  Symptoms of health anxiety are measured by a very short version of a well established patient-rated scale and has been created by factor analytic item-reduction and sensitivity to change analyses from large datasets from previous trial within the research group. The scale ranges from 0 to 9 points. A lower score means less symptoms of health anxiety. As such, a lower score is a better outcome.
Obsessive Compulsive Disorder 3-Item (OCD-3-MINI) | Change during the period Pre-Week4-Week8-Week 52
  Symptoms of obsessive compulsive disorder are measured by a very short patient-rated scale and has been created by an expert group. The scale ranges from 0 to 12 points. A lower score means less obsessive/compulsive thoughts and behaviors. As such, a lower score is a better outcome.
Pain One-item Rating | Change during the period Pre-Week4-Week8-Week 52
  Pain is measured on a scale from 0 to 10, where 0 is no pain and 10 is worst pain imaginable. As such, a lower score is a better outcome.
Total symptom index | Change during the period Pre-Week4-Week8-Week 52
  Also, a total index for level of symptoms will be calculated from all 21 symptom items, where different weights will be used to balance the different number of questions for different domains, for example to avoid the larger number of items related to anxiety to overshadow depression ratings. The scale ranges from 0 to 20 points. A lower score means less mental health symptoms overall. As such, a lower score is a better outcome.
Brunnsviken Brief Quality of Life Questionnaire | Change during the period Pre-Week4-Week8-Week 52
  Quality of life will be measure be the 12-item Brunnsviken Brief Quality of life (BBQ-12), asking about importance and fulfilment of six areas (e.g. spare time quality, creative work, and friendship). The scale ranges from 0 to 96 points. A lower score means lower quality of life. As such, a higher score is a better outcome.
Patient-rated problem severity, Confidence in ability to change, and Helpfulness of visit | Change from visit to visit through study completion (average of 8 weeks)
  All rated from 1-10 by patient when asked by clinician. A lower score means lower symptoms / confidence / helpfulness. As such, a lower score is a better outcome for the symptom question but a worse outcome for the confidence and helpfulness questions.
  Questions are administered at every visit. There is no set time frames as visits can have irregular spacing and different participants will have varying numbers of visits. These questions do not make up a validated scale, but are clinically used within Focused Acceptance and Commitment Therapy.
One item Clinical Global Impression - Improvement (CGI-I) | 4 weeks, 8 weeks
  Related to main problem seeking care for as rated by clinician. The scale ranges from 0 to 7 points. A lower score means a larger improvement for the patient. As such, a lower score is a better outcome.
Patient-rated perception and attitude toward care provider | 4 weeks, 8 weeks
  9-items previously used in PCBH-settings (self-report), and four items from the Client Satisfaction Questionnaire (CSQ). The scale ranges from 0 to 57 points. A lower score means less satisfaction with care. As such, a higher score is a better outcome.
Description of Behavioral Health Plan (PCBH) or main treatment goal and methods (shCBT) as structured note by clinician in medical record | 4 weeks, 8 weeks, 52 weeks
  Interview form.
Patient recollection of plan/goal/methods, descriptions of behaviour changes made | 4 weeks, 8 weeks, 52 weeks
  Interview form.
Experienced negative/Adverse Events, where the worst and most probably care-induced event is more thoroughly described and rated on severity and perceived cause | 4 weeks, 8 weeks, 52 weeks
  Interview form.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, Professor, Principal Investigator — Linnaeus University
Locations (2):
- Sweden (2):
  - Vårdcentralen Centrum, Vaxjo, Kronoberg County
  - Capio Citykliniken Västra Hamnen, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No